CLINICAL TRIAL: NCT02256735
Title: A Double-blinded, Randomised, Placebo Controlled, Five-way Crossover Study With One Positive Control (Open-label) (Moxifloxacin) to Assess the Influence of Oral Single Dose KUC 7483 BS (40 mg, 80 mg, 160 mg, 320 mg) on the QT/QTc Interval of the ECG in Healthy Male and Female Volunteers
Brief Title: Study to Investigate the Effect of KUC 7483 CL on the QT/QTc Interval of the ECG in Comparison to Placebo and Moxifloxacin in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1207.22
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Culture Media; Moxifloxacin

ARMS (6):
- Treatment A (Experimental)
  Interventions: Drug: Treatment A
- Treatment B (Experimental)
  Interventions: Drug: Treatment B
- Treatment C (Experimental)
  Interventions: Drug: Treatment C
- Treatment D (Experimental)
  Interventions: Drug: Treatment D
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Treatment A — Ritobegron Cl (KUC 7483 CL) tablets low dose
  Arms: Treatment A
Drug: Treatment B
  Other Names: Ritobegron Cl (KUC 7483 CL) tablets medium 1 dose
  Arms: Treatment B
Drug: Treatment C
  Other Names: Ritobegron Cl (KUC 7483 CL) tablets medium 2 dose
  Arms: Treatment C
Drug: Treatment D
  Other Names: Ritobegron Cl (KUC 7483 CL) tablets high dose
  Arms: Treatment D
Drug: Placebo
  Arms: Placebo
Drug: Moxifloxacin
  Arms: Moxifloxacin

SUMMARY:
Study to investigate the effect of Ritobegron CL (KUC 7483 CL) on the QT/QTc interval of the ECG in comparison to placebo and moxifloxacin

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females
* Age 30 to 60 years
* Body mass index (BMI) within 18.5 to 29.9 kg/m2
* In accordance with Good Clinical Practice (GCP) and the local legislation all volunteers are to have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, clinically relevant electrolyte disturbances
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or clinically relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (within two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Drug abuse
* Blood donation (> 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the reference range if indicative of underlying disease or poor health
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to treatment medication, moxifloxacin and/or related drugs of these classes
* Previous tendon disease related to quinolone treatment
* Congenital or documented acquired QT- prolongation, previous history of symptomatic arrhythmias
* Heart rate at screening of > 80 bpm or < 45 bpm
* Any screening ECG value outside of the reference range of clinical relevance including, but not limited to Pulse rate (PR) interval > 220 ms, QRS interval > 115 ms, QTcB > 450 ms, or QT (uncorrected) > 470 ms

For Female Subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception e.g. sterilization, Intrauterine pessary (IUP), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2005-08; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean time-matched QTcI | up to 2 hours following drug administration

SECONDARY OUTCOMES:
Change from baseline in mean time-matched QTcI | up to 8 hours following drug administration
Occurrence of uncorrected QT interval | up to 8 hours following drug administration
  QT interval <=500 ms, > 500 ms
Occurrence of the QTcI interval | up to 8 hours following drug administration
  QTcI interval <= 450 ms, >450 ms, >480 ms or >500 ms
Change from baseline of the QTcI interval | up to 8 hours following drug administration
  QTcI interval < 30 ms, ≤ 60 ms
Change from baseline in Heart Rate (HR) | up to 6 hours following drug administration
  increase ≥25 % or decrease HR by ≥25 %
Cmax (maximum measured concentration of the analyte in plasma) | up to 8 hours following drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 8 hours following drug administration
AUC0-6 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 6 hours) | up to 6 hours following drug administration
AUC0-8 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 8 hours) for moxifloxacin | up to 8 hours following drug administration
Number of subjects with adverse events | up to 17 days after last drug administration
Number of subjects with abnormal changes in laboratory parameters | up to 17 days after last drug administration
Number of subjects with abnormal changes in 12-lead ECG | up to 17 days after last drug administration
Number of patients with clinically significant changes in vital signs | up to 17 days after last drug administration
  Blood pressure, pulse rate
Assessment of tolerability by investigator on a 4-point scale | 17 days after last drug administration